CLINICAL TRIAL: NCT02570828
Title: Thermal Imaging in Neonates: a Feasibility Study in Healthy Babies and Babies With Suspected Transient Tachypnea of the Newborn (TTN)
Brief Title: Thermal Imaging in Neonates: A Feasibility Study in Healthy Babies and Babies With Suspected TTN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief, Division of Global Health, Department of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015P001500
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Thermal Imaging, Neonatal Pneumonia, Tachypnea
Keywords: healthy neonate, tachypnea, thermal imaging, pneumonia
MeSH Terms: conditions — Tachypnea; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermal imaging (Experimental): All subjects in the study will have thermal images of the chest taken using the FLIR ONE attachment to an iPhone.
  Interventions: Device: Thermal Imaging

INTERVENTIONS:
Device: Thermal Imaging — FLIR ONE attachment to an iPhone

SUMMARY:
This is a study to evaluate thermal imaging as a technology to monitor the normal clearing of amniotic fluid from healthy newborns and newborns suspected of having a condition called transient tachypnea of the newborn, or TTN. Thermal images are taken using an imaging device that attaches to an iPhone. This device, commercially known as FLIR ONE, creates a non-identifiable image based on the heat pattern of an object. In this case, the object is a child's chest and back. It does not emit any radiation like an x-ray does.

ELIGIBILITY:
Inclusion Criteria (healthy and suspected TTN babies):

* Full term (greater than or equal to 37 weeks gestation)
* less than 3 days old
* born via normal vaginal delivery

Inclusion Criteria (only for suspected TTN babies):

* neonatologist assesses baby as possibly having TTN
* chest x-ray done as part of evaluation for TTN
* no other significant co-morbid conditions present

Exclusion Criteria:

* parents do not consent to have baby participate

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
asymmetric heat distribution | within the first 3 days of life
  thermal imaging will be used to capture asymmetric heat distribution across lung fields

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States